CLINICAL TRIAL: NCT00561444
Title: A Comprehensive, Multimodality Quality of Life Study for Prostate Cancer Patients
Brief Title: Quality of Life Study for Prostate Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0302
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Radical retropubic prostatectomy; Robotic prostatectomy; Photon external beam radiation; Photon external beam radiation with hormone therapy; Proton radiation; Radioisotopic implant; Cryotherapy; Quality of Life; Questionnaire; Survey; QOL
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Quality of Life Study: Prostate cancer patients
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires taking 20 minutes to complete.
  Other Names: Survey

SUMMARY:
The goal of this behavioral research study is to look at patients' quality of life after treatment or management for prostate cancer.

DETAILED DESCRIPTION:
Questionnaires:

You will complete 2 questionnaires that will ask you questions about your quality of life, urinary, bowel, sexual function, and any side effects that you may be having. You will be asked about any medications you may be taking and any other medical conditions you may have. The questionnaires will take about 20 minutes to complete. You may complete the questionnaires at the clinic, have them mailed to you (return postage will be included), or be asked the questions over the phone.

If you are on active surveillance (checking for prostate cancer by routine blood draws and biopsy, without active treatment), you will fill out the questionnaires on the same schedule as those receiving treatment that does not involve hormones.

If you are receiving therapy that does not involve hormones, you will complete the questionnaires before you receive treatment.

If you are receiving hormone therapy, you will complete the questionnaires before beginning the hormone therapy and then again within 3 weeks before starting radiation.

For all participants, at 3 and 6 months after the treatment is completed, you will complete the questionnaires again. Starting 6 months after you finish treatment, you will complete the questionnaires every 6 months for 2 years. Starting 2 years after treatment, you will complete the questionnaires once a year for 3 years.

Length of Study:

All participants will be considered off-study once they have completed the last questionnaires. You will be taken off study early if you receive a second treatment for prostate cancer or if you decide to have treatment while on active surveillance.

This is an investigational study. Up to 1448 patients will be enrolled in this study. All will be enrolled at MD Anderson, MD Anderson Albuquerque, and MD Anderson Cooper.

ELIGIBILITY:
Inclusion Criteria:

1. Primary treatment at MD Anderson for prostate cancer using: radical retropubic prostatectomy, robotic prostatectomy, photon external beam radiation, photon external beam radiation with hormone therapy, proton radiation, radioisotopic implant, cryotherapy, or active surveillance.
2. Neoadjuvant, concurrent and adjuvant androgen ablation in conjunction with photon external beam radiation is allowed if not greater than 6 months total duration. Hormone therapy will be given as an LHRH agonist with or without an antiandrogen.
3. Pathologic diagnosis of prostate adenocarcinoma
4. AJCC (VI) stage T1-T3b N0M0
5. Ability to read, write, and fill out the self-survey questionnaires
6. Patients may be simultaneously enrolled on other MD Anderson treatment or laboratory protocols. The EPIC Survey will be used for both this protocol and for protocol 2007-0209 such that patients enrolled on both protocols will complete only one document at each survey point. Simultaneous enrollment on other survey protocols will be handled in a similar manner.

Exclusion Criteria:

1. Histology other than adenocarcinoma
2. Stage T4, nodal or distant metastasis
3. Prior treatment for prostate cancer except for neoadjuvant, concurrent and adjuvant androgen deprivation of 6 months or less duration in patients treated with photon radiation. Hormone therapy in all other modalities is not allowed.
4. Chemotherapy or molecular targeting therapy as primary, neoadjuvant or adjuvant treatment
5. Treatment for another pelvic malignancy, to include surgery or radiation
6. Treatment for another malignancy with chemotherapy completed within one year or less of treatment for prostate cancer.
7. Inflammatory bowel disease (eg. Crohn's or Ulcerative Colitis)
8. Patients 18 years or younger.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1051 (Actual)
Dates: Start 2007-11-14 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
QOL: Expanded Prostate Cancer Index Composite (EPIC) Survey | Survey prior to beginning treatment, 3 months after completing treatment, 6 months after completing treatment, at 6 month intervals for the first 2 years post-treatment, and then yearly for 3 more years.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A. Kuban, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - MD Anderson at Cooper, Voorhees Township, New Jersey
  - MD Anderson Cancer Center at Albuquerque, Albuquerque, New Mexico
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org